CLINICAL TRIAL: NCT00607880
Title: A Prospective Randomized Study of the Vortex® Implantable Access Port Versus the BardPort™ Implantable Port in Cancer Patients Receiving Adjuvant Intravenous Chemotherapy
Brief Title: Study Comparing Two Types of Ports in Patients With Cancer Receiving Intravenous Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P30CA015083 (NIH); P30CA015083 (NIH); 52-04 (Other: Mayo Clinic Cancer Center & Mayo Clinic IRB)
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Vascular Access Device Complications
Keywords: vascular access device complications; unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Port (Active Comparator): Patients undergo insertion of the conventional vascular access port (C. R. Bard, Inc., Murray Hill, NJ). Patients then receive standard chemotherapy.
  Interventions: Procedure: vascular access device placement
- Vortex Implantable Access Port (Experimental): Patients undergo insertion of the Vortex® implantable vascular access port (Horizon Medical Products, Manchester, GA). Patients then receive standard chemotherapy.
  Interventions: Procedure: vascular access device placement

INTERVENTIONS:
Procedure: vascular access device placement

SUMMARY:
RATIONALE: Giving chemotherapy drugs through an implanted port reduces the need for multiple needle sticks. It is not yet known whether one type of port is more effective than another in reducing infections and other side effects associated with long-term port use.

PURPOSE: This randomized clinical trial is comparing two types of ports in patients with cancer receiving intravenous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the rate of port failure, defined as the occurrence of port malfunction or port infection within 12 months after port insertion, in patients with cancer requiring long-term adjuvant intravenous chemotherapy undergoing insertion of a newly designed, FDA-approved Vortex® implantable vascular access port vs a conventional vascular access port.

Secondary

* To compare the rate of port malfunction or port infection at 6 and 12 months after port insertion.
* To compare the rate of central vein thrombosis at 6 and 12 months after port insertion.
* To compare the rate of port removal for any reason other than infection or occlusion at 6 and 12 months after port insertion.
* To compare the rate of termination of use of the indwelling port at 6 and 12 months after port insertion.
* To compare the death from all causes.
* To compare the incidence of port-related interventions at 6 and 12 months after port insertion.

OUTLINE: Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo insertion of a conventional vascular access port. Patients then receive standard chemotherapy.
* Arm II : Patients undergo insertion of the Vortex® implantable vascular access port. Patients then receive standard chemotherapy.

All episodes of access to the port are documented for 12 months after port insertion. Information including the reason for port access and difficulty in access is collected. Complications, such as occlusion and infection, implant duration, and incidence of port-related interventions are assessed at 6 and 12 months after port insertion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignancy requiring intravenous chemotherapy for ≥ 6 months

  * Must undergo entire course of chemotherapy at the Mayo Clinic in Jacksonville, unless the outside treating institution agrees to submit the research data sheet to Mayo Clinic
* Scheduled time frame for regular use of the vascular access port ≥ 3 months after port insertion

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* No active skin condition implicating an elevated risk of local or systemic infectious or non-infectious complications, including any of the following:

  * Current skin infection
  * Cutaneous lymphoma
  * Auto-immune disorders
  * Active vasculitis
  * Connective tissue diseases
* No known active infection requiring antibiotic therapy at the time of port implantation

  * Patients without an active infection who are on chronic antibiotic suppressive therapy are eligible
* No concurrent illness requiring chronic anticoagulation

  * Patients who develop other comorbidities requiring chronic anticoagulation during the study period are eligible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert G. Hakaim, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Jacksonville, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients considered for port implantation for intravenous chemotherapy were consulted and evaluated for port implantation. This evaluation was not study specific. If the implantation of a port system was feasible, the patient fulfilled inclusion criteria and the patient consented to the study, then they were randomly assigned a treatment port.
Pre-assignment Details: One patient in the Standard Access Port group was unable to have the port placed due to chronic left internal jugular occlusion and was excluded from the analyses.
Groups:
- Standard Access Port: Patients undergo insertion of the conventional vascular access port (C. R. Bard, Inc., Murray Hill, NJ). Patients then receive standard chemotherapy.
Period: Overall Study
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0
Not completed — Unable to place port due to occlusion | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 100 patients accrued to participate in this study were included in the baseline population analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Access Port | Vortex Implantable Access Port | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 93] | 64 [31 to 81] | 65 [31 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Port Failure Within 12 Months of Port Insertion
Description: We report the proportion of patients in each treatment group who have some degree of port failure. Port failure is defined as the composite outcome of port malfunction due to partial or total occlusion and any infection related to the port, within 12 months of port insertion. The percentages reported here are the number of patients that had reported a port failure within 12 months out of the number of patients with port failure within 12 months plus the number of patients that were followed 12 months without port failure.
Time Frame: Up to 12 months from port insertion
Population: Patients with port failure within 12 months and patients that were followed 12 months without port failure were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Number analyzed (Participants) | 31 | 29
percentage of patients | 16.1 [3.2 to 29.0] | 13.8 [1.2 to 26.4]

2. Secondary Outcome: Death From All Causes
Description: Number of patients that died during treatment due to any cause.
Time Frame: Up to 12 months after port insertion
Measure: Number; unit: participants
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Number analyzed (Participants) | 49 | 50
participants | 9 | 6

3. Secondary Outcome: Port Removal for Any Reason Other Than Infection or Occlusion Within 12 Months After Port Insertion
Description: We report the number of patients that terminated use of port due to any reason other than infection or occlusion within 12 months.
Time Frame: Up to 12 months after port insertion
Population: All patients accrued to this study that had their port removed within12 months for any reason other than infection/occlusion were included in this analysis. 28 patients using the Standard Access Port and 30 patients using the Vortex Implantable Access Port had port removal prior to 12 months due to reasons other than infection or occlusion..
Measure: Number; unit: participants
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Number analyzed (Participants) | 28 | 30
participants
  Death | 9 | 6
  End of Chemotherapy | 7 | 6
  Skin Erosion | 1 | 0
  Unhealed Incision | 1 | 0
  Thrombosis | 0 | 1
  Patient Moved/Transferred Care | 4 | 7
  Patient Request | 1 | 0
  Unknown | 5 | 10

4. Secondary Outcome: Termination of Use of the Indwelling Port at 12 Months After Port Insertion
Description: The number of patients that discontinued use of inserted port for any reason at the 12 month timepoint.
Time Frame: Up to 12 months after port insertion
Measure: Number; unit: participants
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Number analyzed (Participants) | 49 | 50
participants | 31 | 31

ADVERSE EVENTS:
Arm/Group | Standard Access Port | Vortex Implantable Access Port
Serious Adverse Events (participants affected / at risk) | 5/49 | 4/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Access Port (N=49) | Vortex Implantable Access Port (N=50)
Vascular - Other (Vascular disorders) | 4 (4) | 2 (2) — Vascular Access Complication, Port Occlusion
Infection with unknown ANC: Blood (Infections and infestations) | 2 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No